CLINICAL TRIAL: NCT07333846
Title: Development of a Landmark-formula for Distal Cephalic Vein Localization and Validation Study of Accuracy in Pediatric Patients
Brief Title: A New Landmark-formula for Cephalic Vein in Children
Status: Recruiting | Type: Observational
Sponsor: Alexander Schmidt (Other)
Responsible Party: Sponsor-Investigator, Alexander Schmidt, Vice Chief Department of Pediatric Anesthesia & Program Director for Research and Education, University Children's Hospital Zurich, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Other Study IDs: KEK-ZH-Nr.: 2025-01 980
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Venipuncture; Ultrasound; Difficult Intravenous Access in Pediatrics; Pediatric Anesthesia
Keywords: landmark; peripheral venous access; cephalic vein; vena cephalica; ultrasound-guided venipuncture; ultrasound-guided placement intravenous line

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In children undergoing surgery, a venous access line almost always has to be placed. Through this line, medications and fluids can be administered during anesthesia or later during the hospital stay. In young children, it is often difficult to find a suitable vein. This can lead to multiple puncture attempts and may be a traumatic experience for both children and their parents. With ultrasound, however, in such difficult cases a specific vein on the forearm (the "cephalic vein") can usually be visualized and cannulated. Mostly, this vein is not visible to the naked eye.

In our research project, we aim to determine whether it is possible to identify a simple and reliable anatomical orientation aid ("landmark") on the forearm that enables parents to place a topical anesthetic EMLA patch precisely at the correct location where the vein can subsequently be found using ultrasound. In this way, we want to assess whether this method simplifies the preparation for venipuncture and thereby increases the success rate. The examination is carried out during the routine preparation for anesthesia.

In a first step, the course of the vein is identified by ultrasound, marked on the skin in a controlled manner, and photographic documentation of the forearm region is created. From this, a visual orientation guide describing the landmark is developed. In a second step, parents and staff of the anesthesia department mark the defined landmark using this visual orientation guide. Ultrasound is then used again to verify whether the vein is located at the marked site. No additional needle puncture is performed and no additional blood sample is taken.

DETAILED DESCRIPTION:
This study is a prospective, single-center, observational validation study designed to develop and evaluate a reproducible external anatomical landmark for localization of the distal cephalic vein at the forearm in pediatric patients. The study aims to support accurate preprocedural placement of topical local anesthetic (EMLA) and to facilitate subsequent peripheral venous access in children by using ultrasound as the reference standard.

Background and Rationale

Peripheral venous access in young children is frequently challenging due to limited visibility and palpability of superficial veins. The cephalic vein at the distal forearm is a commonly used site for ultrasound-guided cannulation; however, standardized external anatomical landmarks for preprocedural localization of this vein are lacking, particularly in pediatric patients. As a result, opportunities for timely application of topical anesthetics are often missed, especially in ambulatory and day-surgery settings where parents are required to apply EMLA patches at home prior to hospital admission.

Ultrasound provides accurate visualization of superficial venous anatomy and allows objective validation of surface landmark accuracy. This study seeks to define a practical, reproducible landmark for the distal cephalic vein and to assess whether this landmark can be applied reliably by anesthesia professionals as well as by parents or caregivers using a standardized visual instruction guide.

Study Design and Setting

The study is conducted at a single Swiss university children's hospital and consists of two sequential, non-interventional study parts. All ultrasound examinations are performed intraoperatively after induction of general anesthesia for clinically indicated elective surgery. No venipuncture or deviation from standard clinical care is performed as part of the study.

Each participant contributes data at a single time point only. No follow-up visits or longitudinal assessments are planned.

Study Procedures

Study Part 1 - Pilot Phase (Landmark Development):

In an initial pilot phase, ultrasound examinations of the distal cephalic vein are performed in a cohort of pediatric patients under general anesthesia. The vein's course, depth, and diameter are assessed, and the vein's trajectory is marked on the skin with a washable marker. Photographic documentation of the forearm is obtained. Based on these sonographic measurements and images, a reproducible external anatomical landmark is developed for use in the validation phase.

Study Part 2 - Validation Phase:

The predefined anatomical landmark is evaluated in two independent validation steps:

Step 1 (Anesthesia Staff Application):

Anesthesia professionals apply the landmark by marking the presumed vein location on the forearm using a washable marker, guided by a standardized visual instruction. After induction of anesthesia, ultrasound is used to determine whether the cephalic vein is located beneath the marked area and to document anatomical parameters.

Step 2 (Parent/Caregiver Application):

Parents or caregivers apply an EMLA patch to the forearm using the same visual instruction guide prior to surgery. After induction of anesthesia, the patch is removed and ultrasound examination is performed to assess whether the cephalic vein is located beneath the area covered by the patch.

In both validation steps, ultrasound measurements are performed by anesthesia personnel not involved in the initial marking to reduce observer bias.

Ultrasound Assessment

Ultrasound examinations are performed using high-frequency linear probes suitable for pediatric vascular imaging. The following parameters are documented at the marked site:

* Presence of the cephalic vein within the marked or EMLA-covered area
* Distance between the center of the vein and the center of the marked area
* Vein depth from the skin surface
* Vein diameter
* Proximal course of the vein over a distance of up to 3 cm

All measurements are obtained with the patient under general anesthesia to avoid movement-related variability.

Data Collection and Management

Study data are recorded using standardized paper Case Report Forms (CRFs) and subsequently transferred to a secured electronic database. Data are pseudonymized at the time of collection. Ultrasound images and photographic documentation are stored digitally to allow verification if required.

Source data include CRFs, ultrasound images, and relevant routine clinical data (e.g., age, weight). No biological samples are collected, and no questionnaires or laboratory tests are performed.

Quality Assurance and Monitoring

Several measures are implemented to ensure data quality and consistency:

* Standardized ultrasound procedures and documentation checklists
* Training and briefing of all participating sonographers
* Use of standardized visual instruction guides for landmark application
* Partial double data entry and random data checks
* Internal monitoring by the principal investigator
* Secure storage and version control of all study documents
* The study may be subject to audits or inspections by the responsible ethics committee, with direct access to source data if required.

Sample Size Considerations

This is an exploratory, non-confirmatory study. A formal power calculation was not performed. The planned sample size for the validation phase is based on achieving sufficient precision in estimating the proportion of correctly localized veins. Inclusion of approximately 30 participants per validation subgroup allows estimation of the primary accuracy measure with acceptable confidence interval width for an exploratory anatomical validation study.

Statistical Analysis Principles

Data analysis is primarily descriptive. Continuous variables are summarized using measures of central tendency and dispersion, while categorical variables are summarized using proportions and confidence intervals. Exploratory analyses assess relationships between anatomical parameters and demographic variables such as age, body weight, and body mass index. No interim analyses are planned.

Handling of Missing Data

Missing data may occur due to technical limitations or incomplete documentation. Analyses are performed using available data only, without imputation. If the number of evaluable cases falls below predefined targets, recruitment may be extended to ensure adequate data completeness.

Ethical and Safety Considerations

The study involves minimal risk. All procedures are non-invasive and performed under general anesthesia as part of routine clinical care. No additional pain, radiation exposure, or biological sampling is involved. Data protection measures include pseudonymization during data collection and anonymization after completion of the analysis. The study is conducted in accordance with applicable ethical and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Children under the age of 6 years
* Scheduled elective procedure under general anesthesia
* Admission via the surgical day clinic
* Written informed consent by the parents (and by the child if capable of judgment)

Exclusion Criteria:

* pre-existing intravenous access at the investigation site
* Skin conditions or infections at the forearm site
* Known allergy to EMLA or any of its components

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children under 6 years of age scheduled for elective surgery under general anaesthesia at a single tertiary paediatric centre in Switzerland. Participants are recruited consecutively from the preoperative surgical list; parent/guardian consent is obtained. Setting: Department of Anaesthesiology, University Children's Hospital, Zurich, Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Hit rate of cephalic vein within the marked and EMLA-covered area | Baseline (one ultrasound-examination after induction of anesthesia for planned surgery)
  Proportion of cases where the cephalic vein is found within the user-marked area (staff or parent) and covered by the EMLA patch. (binary: yes/no). All outcome measures are assessed by ultrasound under general anesthesia.

SECONDARY OUTCOMES:
Distance (mm) | Baseline (one ultrasound-examination after induction of anesthesia for planned surgery)
  Distance (mm) between vein center and center of marked area
Vessel diameter (mm) | Baseline (one ultrasound-examination after induction of anesthesia for planned surgery)
  Maximal vessel diameter (mm) at the marked location in transverse plane during venostasis
Vessel depth (mm) | Baseline (one ultrasound-examination after induction of anesthesia for planned surgery)
  Vessel depth (mm) from skin surface to vein center
Proximal course of the vein | Baseline (one ultrasound-examination after induction of anesthesia for planned surgery)
  Proximal course of the vein, defined as visibility and continuity of the vein over a 3 cm proximal segment (categorical: straight / curved / splitting up)
Correlation of venous anatomy and patient characteristics | Baseline (one ultrasound-examination after induction of anesthesia for planned surgery)
  Correlation of venous depth and diameter with age, weight and BMI
Feasibility comparison | Baseline (one ultrasound-examination after induction of anesthesia for planned surgery)
  Feasibility comparison between marking performed by anesthesia personnel and by parents, measured as difference in hit rate

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Schmidt, MD, Study Chair — University Children's Hospital, Zurich
Locations (1):
- University Childrens Hospital, Department of Anaesthesia and Children's Research Centre, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. De-identified data may be transmitted to the journal/publisher to meet publication requirements. Any further use of participant-level data outside this study is excluded by protocol and consent. Aggregate results and analysis methods will be available in publications